CLINICAL TRIAL: NCT03530748
Title: On-table Renal Perfusion Evaluation for Patients With Renal Artery Stenosis or Aortic Dissection With Renal Artery Obstruction
Brief Title: On-table Renal Perfusion Evaluation Renal Artery Stenosis or Obstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Zhenyu Shi, Clinical Professor, Shanghai Zhongshan Hospital
Other Study IDs: B2017-084
Record Dates: First submitted 2018-04-10; First posted 2018-05-21 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Renal Artery Stenosis; Aortic Dissection; Renal Perfusion; Renal Artery Obstruction
MeSH Terms: conditions — Renal Artery Obstruction; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Renal Artery Stenosis: Patients with simple renal artery stenosis or aortic dissection with renal artery obstruction
  Interventions: Procedure: Endovascular therapy and Imaging Acquisition

INTERVENTIONS:
Procedure: Endovascular therapy and Imaging Acquisition — 1. Endovascular repair for renal artery stenosis;
  2. Parenchymal Blood Volume(PBV) acquisition and analysis for target kidney

SUMMARY:
1. Evaluate the feasibility for the on-table evaluation of the renal perfusion by using Syngo Dyna Parenchymal Blood Volume(PBV) Body;
2. Explore the clinical benefits of this application during procedure to help the physician to determine the procedure endpoint.

DETAILED DESCRIPTION:
Renal artery stenosis (RAS) is one of the potential manifestations of peripheral artery diseases and it is often observed in patients with evolving renal function impairment and concomitant coronary artery disease, or in those suffering from hypertension refractory to medical therapy.Percutaneous renal artery stenting is an effective therapeutic tool and represents the treatment of choice for RAS. Identification of parameters able to discriminate patients who benefit from RAS stenting, thus, has become of crucial importance if this technique has to survive.

Aortic dissection represents a common cardiovascular disease and it is responsible for the most commonly encountered pathologies in aortic emergency. Renal dysfunction is a common complication associated with aortic dissection, with resultant high mortality rate. The antegrade propagation of the dissection from the proximal aorta to the level of renal arteries and the intervention during surgery may both increase the risk of renal malperfusion; thus, it is important to assess renal function for pre- and post-operative evaluation and guidance for treatment. This can be achieved through perfusion imaging.

Presently, C-arm Cone Beam Computed Tomography (CBCT) perfusion is well established, in particular, in the diagnostic assessment of acute stroke and cerebral ischemia. The main novelty of our study lies in the fact that intra-procedural renal perfusion assessed for the first time semiquantitatively by Syngo Dyna Parenchymal Blood Volume(PBV) software, discriminate patients who will benefit from the intervention procedure.

In conclusion, our study suggests that a routine assessment of pre, and post-stenting renal perfusion could help to identify patients at higher risk of no improvement or even worsening of renal function after stenting and, perhaps, more aggressive medical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Renal artery stenosis ≥ 60% and < 100% by doppler ultrasonography, CT angiography or magnetic resonance angiography;
* Target kidney remains functional (GFR determined);
* The length of target kidney is >8cm;
* Resistance index tested by doppler ultrasonography <0.8;
* Comply with the protocol

Exclusion Criteria:

* Severe cardiopulmonary insufficiency, hepatic dysfunction, renal inadequacy and clotting mechanism abnormality;
* Pregnancy or lactation;
* History of renal artery surgery;
* Allergy of contrast agent;
* Other known reason nonischemic kidney disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who meet the inclusion criteria, are willing to comply with this protocol, and receive endovasculara therapy in the Department of Vascular Surgery, Zhongshan Hospital will be included.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-06-09 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate | Change from Baseline Glomerular Filtration Rate at 3 months
  The golden standard of renal function, tested by radionuclide imaging

SECONDARY OUTCOMES:
Kidney Volume | 10 minutes pre- and post-endovascular therapy on table
  Total blood volume of kidney, tested by PBV
Mean Density of Contrast agent | 10 minutes pre- and post-endovascular therapy on table
  Renal blood perfusion, tested by PBV

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Shi, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No